CLINICAL TRIAL: NCT01745029
Title: Gastrointestinal Motility in Patients Suffering From Severe Ulcerative Colitis Obtained by Motilis-3D-transit
Brief Title: Gastrointestinal Motility in Severe Ulcerative Colitis Obtained by Motilis-3D-transit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Motilis Medica A/S ,Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012013250
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Ulcerative Colitis
Keywords: Gastrointestinal Motility; Inflammatory Bowel Disease; Transit time
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ulcerative Colitis
  Interventions: Device: Motilis-3D-transit

INTERVENTIONS:
Device: Motilis-3D-transit

SUMMARY:
The purpose of this study is to describe gastrointestinal (GI) motility in patients suffering from severe Ulcerative Colitis (UC) and to compare these results with similar results obtained in remission.

The study is done with the use of Motilis 3D-Transit system which consists of a small electronic capsule ingested and detected by a receiver carried by the patient. Position and orientation of the capsule are interpreted by dedicated computer software and transit times, progression velocity and contraction frequencies can be revealed.

The study is mainly descriptive and is designed to test and evaluate the usefulness of the Motilis 3D Transit system in UC patients and to tell investigators more about GI motility during and after severe inflammation.

Motilis 3D-Transit system gives investigators a unique chance to study the gastrointestinal canal as a whole during and after severe illness.

The investigators expect to include 20 patients suffering from severe UC admitted to Hospital with the purpose of getting medical treatment. The investigators do not expect any drop out, but in case of drop out a new patient will be included.

ELIGIBILITY:
Inclusion criteria:

* Severe Ulcerative colitis (modified Truelove and Witt score)
* Signed informed consent obtained
* Fasted since midnight

Exclusion Criteria:

* Known GI related symptoms complaints or GI diseases
* Swallowing disorders
* Cancer or other life threatening diseases or conditions
* Pregnancy or breast-feeding
* Previous abdominal surgery
* Abdominal diameter >140cm?
* Drug abuse or alcoholism
* Irregular bowel movements
* Known cardiovascular or pulmonary diseases
* Participation in any clinical study within the last 30 days
* Cardiac pacemaker or infusion pump or any other implanted or portable electro-mechanical medical device.
* Medication affecting GI motility
* MRI within the next four weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe Ulcerative Colitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Velocity of progression through the inflamed part of the colon in severe UC compared to the velocity of progression in the corresponding colonic segment in quiescent UC. | Three days from baseline visit

SECONDARY OUTCOMES:
Velocity of progression through the non-inflamed colonic segments in severe UC compared to the velocity of progression in the corresponding colonic segments in quiescent UC. | Three days from baseline

OTHER OUTCOMES:
Velocity of progression through the colonic segments in quiescent UC compared to the velocity of progression in the corresponding colonic segments in healthy volunteers. | three days from baseline visit

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Hepato and Gastroenterolegy, Aarhus C, Denmark